CLINICAL TRIAL: NCT03342430
Title: Early Dieting in Girls
Brief Title: Early Dieting in Girls: a Longitudinal Cohort Study
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Assistant Professor, Penn State University
Other Study IDs: HD32973
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Eating Behavior; Dietary Habits; Weight, Body
MeSH Terms: conditions — Feeding Behavior; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early Dieting in Girls cohort: A cohort of 197 non-Hispanic white girls, observed from age 5 to age 15 years

SUMMARY:
This longitudinal observational cohort followed the growth and development of non-Hispanic white girls from age 5 to 15 years, with a focus on the development of the controls of food intake.

DETAILED DESCRIPTION:
This longitudinal observational cohort followed the growth and development of non-Hispanic white girls from age 5 to 15 years, with a focus on the development of the controls of food intake. Data was collected biennially from girls and their mothers and fathers. Measures included anthropometrics, questionnaires and laboratory measures of eating behavior, dietary recalls, psychosocial characteristics, and parenting measures.

ELIGIBILITY:
Inclusion Criteria:

* Living with both biological parents

Exclusion Criteria:

* Severe food allergies
* Chronic medical conditions affecting food intake

Ages: 5 Years to 6 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only girls age 5-6 years old at enrollment and their biological parents were eligible for the study.
Study Population: Families in central Pennsylvania with a 5-6 year old daughter.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 1996-06 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Dieting practices | Pattern of development from age 5 to 15 years
  Derived from questionnaire by French et al.
Dietary restraint | Pattern of development from age 5 to 15 years
  Dutch Eating Behavior Questionnaire
Disinhibition | Pattern of development from age 5 to 15 years
  Dutch Eating Behavior Questionnaire
Disordered eating | Pattern of development from age 5 to 15 years
  Children's Eating Attitudes Test/Eating Attitudes Test

SECONDARY OUTCOMES:
Body mass index | Age 5, 7, 9, 11, 13, and 15 years
  Weight in kg/height in meters squared, converted to z-scores using CDC growth charts
Total body bone mineral content | Age 9, 11, 13, and 15 years
  Dual energy x-ray absorptiometry
Dietary intake | Age 5, 7, 9, 11, 13, and 15 years
  3-24 hour dietary recalls

CONTACTS AND LOCATIONS:
Overall Officials: Leann L Birch, PhD, Principal Investigator — Penn State University (at time study was conducted)

REFERENCES:
- [Derived] Hohman EE, Balantekin KN, Birch LL, Savage JS. Dieting is associated with reduced bone mineral accrual in a longitudinal cohort of girls. BMC Public Health. 2018 Nov 22;18(1):1285. doi: 10.1186/s12889-018-6206-y. PMID 30466435